CLINICAL TRIAL: NCT02258633
Title: A Brief Tailored Family-centered Seatbelt Intervention for Hospitalized Trauma
Brief Title: The Seatbelt Intervention Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Peter Ehrlich, Co-Principal Investigator, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HUM00026025
Record Dates: First submitted 2014-10-02; First posted 2014-10-07 (Estimated); Last update posted 2014-10-07 (Estimated); Status verified 2014-10

CONDITIONS: High Risk Population of Part-time Seatbelt Users

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervener Brief Intervention (IBI) (Experimental): Subjects and parents will complete a Brief Motivational Interview (BMI) incorporating personalized feedback, discussion of choices and changes, and therapist led intervention message relating behavioral change and future goals.
  Interventions: Other: Interactive interview and tailored family centered seatbelt safety intervention
- Enhanced Usual Care (No Intervention): Subjects and parents will receive standard trauma care, plus complete brief questionnaires and receive general safety information.

INTERVENTIONS:
Other: Interactive interview and tailored family centered seatbelt safety intervention
  Arms: Intervener Brief Intervention (IBI)

SUMMARY:
The study will use a randomized controlled design testing the effectiveness of the following intervention: (i) intervener brief intervention (IBI) vs. (ii) Enhanced usual care (EUC). The study will identify children ages 2-14 at a pediatric trauma center. Children and their parents who agree to participate in the study will then complete a screening survey to identify part time seatbelt use. Those who screen positive will complete a more detailed baseline survey and then be randomized to one of two study conditions. At one month, a follow up assessment by telephone will be completed.

ELIGIBILITY:
Inclusion Criteria:

* Children ages 7-14 and their parent or guardian, at a pediatric trauma center
* Child admitted to hospital with diagnosis of injury other than sexual assault and suicide
* Identify as part time seat belt users

Exclusion Criteria:

-

Ages: 7 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200 (Actual)
Dates: Start 2009-03; Primary Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Seat belt use | 1 month
  Follow up telephone assessment on full time seat belt use by parent and child
Seat belt knowledge | 1 month
  Follow up telephone assessment on level of knowledge of seat belt use and risk factors
Attitudes | 1 month
  Follow up telephone assessment of positive attitude, motivation, and self-efficacy regarding safety restraint use.